CLINICAL TRIAL: NCT00547209
Title: Anesthésie Totale Intraveineuse en " Boucle d'Asservissement " guidée Par l'Index Bispectral : Effet de l'Adjonction de Protoxyde d'Azote (Effect of Nitrous Oxide on Intravenous Closed-loop Anesthesia)
Brief Title: Effect of Nitrous Oxide on Intravenous Closed-loop Anesthesia
Acronym: Drone-N2O
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-08
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Anesthesia
MeSH Terms: interventions — Air; Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): ventilation with air and oxygen
  Interventions: Drug: air
- 2 (Experimental): ventilation with nitrous oxide and oxygen
  Interventions: Drug: Nitrous oxide

INTERVENTIONS:
Drug: air — 60% air combined with 40% oxygen for ventilation
  Arms: 1
Drug: Nitrous oxide — 60% nitrous oxide combined with 40% oxygen for ventilation
  Arms: 2

SUMMARY:
The main objective of the study is to analyze the influence of nitrous oxide on propofol and remifentanil requirements.

DETAILED DESCRIPTION:
Nitrous oxide is a widely used anesthetic agent. The mechanism of its central action is not completely understood and its importance is questioned.

Total intravenous anesthesia can be driven by a computer using bispectral index as a controller. Such a system matches anesthetic agent requirements to the needs of each individuum and thus allows an unbiased evaluation of the influence of nitrous oxide. Two groups of patients are compared: one ventilated with a oxygen-air mixture and one with oxygen-nitrous oxide mixture. Anesthesia is provided by a "dual-loop" which adapts propofol and remifentanil target concentrations to maintain a bispectral index between 40 and 60 in both groups.

ELIGIBILITY:
Inclusion Criteria:

* General anaesthesia with controlled ventilation

Exclusion Criteria:

* Age lower than 18 years
* Pregnant woman
* Allergy to the propofol or to a muscle myorelaxant
* Patients receiving a psychotropic treatment
* Presence of a central neurological disorder or a lesion cerebral
* Patients having an anomaly of blood cells count preoperative biological assessment
* Patients having had an anaesthesia in the previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Actual)
Dates: Start 2007-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Measure: influence of nitrous oxide on the automated administration of propofol and remifentanil. | during anesthesia

SECONDARY OUTCOMES:
Measure: consequences of the use of nitrous oxide on the performance of the automated administration system. | during anesthesia
Influence of Gender | during anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hopital Foch, 92150 Suresnes, France
Locations (17):
- Hôpital Erasmes, Brussels, Belgium
- France (15):
  - CHU d'Angers, Angers
  - CH Victor Dupouy, Argenteuil
  - CHU de Besançon, Besançon
  - Clinique Saint Augustin, Bordeaux
  - Hôpital Beaujon, Clichy
  - Centre Hospitalier de Dreux, Dreux
  - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - Institut Paoli-Calmettes, Marseille
  - Centre Hospitalier Territorial Gaston Bourret, Nouméa
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Cochin, Paris
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital Foch, Suresnes
  - Institut Claudius Regaud, Toulouse
  - Hôpital Trousseau, Tours
- La Charite, Berlin, Germany

REFERENCES:
- [Background] Liu N, Chazot T, Genty A, Landais A, Restoux A, McGee K, Laloe PA, Trillat B, Barvais L, Fischler M. Titration of propofol for anesthetic induction and maintenance guided by the bispectral index: closed-loop versus manual control: a prospective, randomized, multicenter study. Anesthesiology. 2006 Apr;104(4):686-95. doi: 10.1097/00000542-200604000-00012. PMID 16571963
- [Background] Karalapillai D, Leslie K, Umranikar A, Bjorksten AR. Nitrous oxide and anesthetic requirement for loss of response to command during propofol anesthesia. Anesth Analg. 2006 Apr;102(4):1088-93. doi: 10.1213/01.ane.0000198672.05639.0a. PMID 16551904
- [Derived] Liu N, Le Guen M, Boichut N, Genty A, Herail T, Schmartz D, Khefif G, Landais A, Bussac JJ, Charmeau A, Baars J, Rehberg B, Tricoche S, Chazot T, Sessler DI, Fischler M. Nitrous oxide does not produce a clinically important sparing effect during closed-loop delivered propofol-remifentanil anaesthesia guided by the bispectral index: a randomized multicentre study. Br J Anaesth. 2014 May;112(5):842-51. doi: 10.1093/bja/aet479. Epub 2014 Jan 31. PMID 24486835